CLINICAL TRIAL: NCT07074028
Title: Characterization and Longitudinal Monitoring of Muscular Phenotype in Patients Admitted to Intensive Care for Sepsis.
Acronym: REAMUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024_CHSB_REAMUS; 2024-A02380-47 (Other: ID RCB)
Record Dates: First submitted 2025-06-19; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Sepsis; Myopathy Critical Illness
Keywords: muscle atrophy; electromyography; Muscle Strength; conditioned medium with human serum
MeSH Terms: conditions — Sepsis; Muscular Atrophy | interventions — Electromyography; Blood Specimen Collection; Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Longitudinal characterization of muscle phenotype in ICU participants with sepsis (Experimental): Through successive visits during and after the ICU stay, the muscle phenotype of participants is determined using non-invasive data collection methods (clinical assessments, ultrasound imaging, and electroneuromyography). Blood samples are harvested to assess the participants' inflammatory status and evaluate organ dysfunction.
  Following the ICU stay, in addition to the previously mentioned data, participants' physical and functional autonomy is assessed. Cognitive impairments and symptoms of anxiety and depression are also recorded, along with their nutritional status.
  Interventions: Diagnostic Test: Medical Research Council sum score (MRC-SS) test; Diagnostic Test: Handgrip test combined with surface electromyography (sEMG); Diagnostic Test: Electrical activity during maximal voluntary contraction of the rectus femoris; Device: Musculoskeletal Ultrasound; Device: Diaphragmatic ultrasound; Biological: blood sampling; Device: Electroneuromyogram; Diagnostic Test: 6-minute walk test; Diagnostic Test: Montreal Cognitive Assessment (MoCA); Behavioral: MNA-SF

INTERVENTIONS:
Diagnostic Test: Medical Research Council sum score (MRC-SS) test — Medical Research Council (MRC)-sumscore evaluates global muscle strength. Manual strength of six muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) is evaluated on both sides using MRC scale
Diagnostic Test: Handgrip test combined with surface electromyography (sEMG) — Handgrip test combined with surface electromyography (sEMG) of the flexor digitorum superficialis
Diagnostic Test: Electrical activity during maximal voluntary contraction of the rectus femoris — Surface EMG amplitude (RMS) during maximal voluntary contraction measured by surface electromyography (sEMG) of the rectus femoris
Device: Musculoskeletal Ultrasound — Measurement of the cross-sectional area (CSA) of the rectus femoris by ultrasound
Device: Diaphragmatic ultrasound — Diaphragmatic ultrasound is a non-invasive technique that allows for sequential assessment of diaphragm mobility (excursion) and contraction (thickening) in mechanically ventilated patients
Biological: blood sampling — Blood samples are collected from a radial or femoral arterial catheter, which is part of the routine care of the patients. These samples are taken with the aim to: 1) describe the inflammatory profile (plasma measurements of CRP, IL-1, IL-6, TNFα, IL-10, fibrinogen, ferritin, cortisol), 2) assess organ dysfunction and calculate the SOFA score (arterial blood gases, lactate levels, liver function tests, complete blood count, and blood electrolyte panel)
Device: Electroneuromyogram — Analysis of peripheral neurogenic and myogenic components involved in intensive care unit-acquired muscle dysfunction through the performance of an electroneuromyogram
Diagnostic Test: 6-minute walk test — The 6-minute walk test (6MWT) is a simple test that requires a quiet, indoor, flat 30-meter course, ideally in a straight rectangular hallway
Diagnostic Test: Montreal Cognitive Assessment (MoCA) — The Montreal Cognitive Assessment (MoCA) is the most sensitive rapid assessment test and assesses cognitive functions most broadly (attention, concentration, executive functions, memory, language, visual-constructive abilities, abstraction, calculation, orientation).
Behavioral: MNA-SF — The MNA-SF (Short Form) is a simplified version that allows us to determine whether the elderly person is well nourished, at risk of malnutrition or malnourished.

SUMMARY:
Approximately 40% of patients develop muscle dysfunction during their stay in intensive care, particularly in the context of sepsis. This dysfunction represents an acquired muscle injury that is secondary to the primary illness that led to ICU admission. It affects both the limb muscles and the respiratory muscles of the thoracic cage. Clinically, this manifests as bilateral and symmetrical muscle weakness in the limbs, and contributes significantly to difficulties in weaning patients off mechanical ventilation.

The loss of muscle mass is directly correlated with the severity of the patient's clinical condition and can reach up to 20% of initial muscle mass within just ten days. This rapid and profound atrophy primarily results from an imbalance between increased muscle protein breakdown (catabolism) and insufficient protein synthesis (anabolism). The consequences of this muscle dysfunction are significant and far-reaching, with a marked negative impact on the overall prognosis.

This condition is associated with longer durations of mechanical ventilation and extended stays in the intensive care unit. Beyond the acute phase, patients often experience persistent reductions in physical performance, leading to long-term functional limitations that impair quality of life. Furthermore, ICU-acquired muscle dysfunction has been linked to increased long-term mortality, with excess deaths reported at both one year and five years following ICU discharge. This risk is especially pronounced when the muscle dysfunction is severe and continues beyond the hospitalization period.

Several risk factors for ICU-acquired muscle dysfunction may be modifiable, opening up the possibility for preventive or therapeutic interventions. Two main factors have been identified as particularly relevant: (1) the duration of immobility and muscular inactivity, and (2) the adequacy of nutritional support, especially regarding amino acid intake, which is critical for maintaining muscle protein synthesis.

In response to these factors, early and active mobilization of ICU patients has become a key component of recommended care, often in conjunction with strategies aimed at minimizing the use of sedative medications. These practices are encouraged by international guidelines, reflecting a growing consensus around the importance of maintaining some level of muscular activity even in critically ill patients. However, despite these recommendations, no definitive evidence has demonstrated a clear improvement in patient outcomes associated with early mobilization.

This lack of clear benefit may stem from multiple factors, including the variability in patient severity across clinical trials and, importantly, the timing of the intervention. The anabolic signals triggered by muscle contraction are only effective if they are strong enough to counterbalance the catabolic signals driven by inflammation, infection, or muscle hypoxia-all of which fluctuate over the course of illness and recovery.

Regarding nutritional interventions, the appropriate timing and quantity of calorie and protein intake necessary to support adequate anabolism and mitigate muscle loss remain controversial. Although amino acids are essential for muscle protein synthesis, current studies have not shown consistent improvements in muscle function based on different nutritional strategies in the ICU setting.

Given the high prevalence of ICU-acquired muscle dysfunction in patients with sepsis, its significant impact on outcomes, and the lack of an effective, evidence-based treatment, there is a pressing need to deepen our scientific understanding of this phenomenon. Improving knowledge in this area could lead to more targeted and effective interventions, ultimately helping to preserve muscle mass and function in critically ill patients and improving both their short- and long-term prognosis.

DETAILED DESCRIPTION:
The care provided to participants enrolled in the study remains unchanged. Standard care is administered. In particular, there are no modifications to routine practices regarding early mobilization, physiotherapy, physical exercise, or nutritional management.

The muscular phenotype of enrolled participants is assessed longitudinally during their ICU stay and after hospital discharge. Several follow-up visits are scheduled:

* Visit 1: Inclusion
* Visit 2: Day 3 (D3)
* Visit 3: Day 7 (D7)
* Visit 4: Day 14 (D14)
* Visit 5: Day 21 (D21)
* Visit 6: Day 28 (D28)
* Visit 7: ICU discharge (may occur before D28)
* Visit 8: Day 90 (D90) - End of study

During these visits, the muscular phenotype is evaluated using non-invasive methods (clinical assessments, ultrasound imaging, and electroneuromyography). Blood samples are collected to determine the inflammatory status of participants and to assess dysfunctions in vital organs.

After the ICU stay, in addition to these data, participants' physical and functional autonomy is documented. Cognitive impairments and symptoms of anxiety and depression are also recorded, along with their nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Participants admitted to ICU with an expected length of stay greater than 7 days.
* Expected duration of invasive mechanical ventilation greater than 48 hours.
* Diagnosis of sepsis upon ICU admission (presence of an infection and a SOFA score ≥ 2, or an increase of ≥ 2 points if organ dysfunction was present prior to infection).
* Informed consent obtained from the participant or from a designated surrogate decision-maker

Exclusion Criteria:

* Pregnant women.
* Participants not affiliated with the national health insurance system.
* Participants under legal protection (guardianship or conservatorship).
* Moribund participants (end-of-life patients).
* Participants with active cancer.
* Participants with chronic neuromuscular disorders or admitted to the ICU for an acute neuromuscular condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
MRC score (Medical Research Council). | From enrollment to the end of the participant's study period (maximum 90 days)
  The MRC score allows for a global assessment of muscle function in ICU patients. An MRC score below 48, measured on day 28 or at ICU discharge (if discharge occurs before day 28), defines ICU-acquired weakness (ICU-AW).

SECONDARY OUTCOMES:
Handgrip test combined with surface electromyography (sEMG) | From enrollment to the end of the participant's study period (maximum 90 days)
  Handgrip test combined with surface electromyography (sEMG) of the flexor digitorum superficialis
Electrical activity during maximal voluntary contraction of the rectus femoris | From enrollment to the end of the participant's study period (maximum 90 days)
  Surface EMG amplitude (RMS) during maximal voluntary contraction measured by surface electromyography (sEMG) of the rectus femoris
Musculoskeletal Ultrasound | From enrollment to the end of the participant's study period (maximum 90 days)
  Measurement of the cross-sectional area (CSA) of the rectus femoris by ultrasound
Diaphragmatic ultrasound | From enrollment to the end of the participant's study period (maximum 90 days)
  Diaphragmatic ultrasound is a non-invasive technique that allows for sequential assessment of diaphragm mobility (excursion) and contraction (thickening) in mechanically ventilated patients
Electroneuromyogram | Only during the last visit of the protocol : 90 days after the inclusion
  Analysis of peripheral neurogenic and myogenic components involved in intensive care unit-acquired muscle dysfunction through the performance of an electroneuromyogram
Plasma concentrations of inflammation-related proteins | From enrollment to the end of the participant's study period (maximum 90 days)
  Blood samples are collected from a radial or femoral arterial catheter, which is part of the routine care of the patients. These samples are taken with the aim to describe the plasma inflammatory profile including CRP, IL-1, IL-6, TNFα, IL-10, fibrinogen, ferritin and cortisol concentrations. All these data are reported in a Outcome Measure results data table.
Organ dysfunction assesment | From enrollment to the end of the participant's study period (maximum 90 days)
  Blood samples are collected from a radial or femoral arterial catheter, which is part of the routine care of the patients. These samples are taken with the aim to assess organ dysfunction and calculate the SOFA score (arterial blood gases, lactate levels, liver function tests, complete blood count, and blood electrolyte panel).
6-minute walk test | Only during the last visit of the protocol : 90 days after the inclusion
  The 6-minute walk test (6MWT) is a simple test that requires a quiet, indoor, flat 30-meter course, ideally in a straight rectangular hallway
Montreal Cognitive Assessment (MoCA) | Only during the last visit of the protocole : 90 days after the inclusion
  The Montreal Cognitive Assessment (MoCA) is the most sensitive rapid assessment test and assesses cognitive functions most broadly (attention, concentration, executive functions, memory, language, visual-constructive abilities, abstraction, calculation, orientation).
MNA-SF | Only during the last visit of the protocol : 90 days after the inclusion
  The MNA-SF (Short Form) is a simplified version that allows us to determine whether the elderly person is well nourished, at risk of malnutrition or malnourished.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Brieuc - Paimpol - Tréguier, Saint-Brieuc, France

IPD SHARING:
Plan to Share IPD: Undecided